CLINICAL TRIAL: NCT04360369
Title: Comparison of Intraocular Pressure Measurements Between Reichert Tono-Vera Tonometer and Goldmann Tonometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reichert, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 16305-TPR-28
Record Dates: First submitted 2020-03-16; First posted 2020-04-24 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Intraocular Pressure; Glaucoma
Keywords: Tonometry, Ocular
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: All study-related tests will be conducted in a single stage, with one clinical visit, to a single clinical center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Goldmann Applanation Tonometer (Active Comparator): Measurement of IOP with Goldmann Applanation Tonometer. All subjects will participate in this arm.
  Interventions: Device: IOP with Goldmann Applanation Tonometer
- ORA G3 and ic100 (Active Comparator): Measurement of IOP with Ocular Response Analyzer G3 and ic100 tonometers. All subjects will participate in this arm.
  Interventions: Device: IOP with comparator ORA G3 and ic100 tonometers
- Tono-Vera Tonometer (Experimental): Measurement of IOP with Tono-Vera Tonometer. All subjects will participate in this arm.
  Interventions: Device: IOP with Tono-Vera Tonometer

INTERVENTIONS:
Device: IOP with Goldmann Applanation Tonometer — Measurement of intraocular pressure (IOP) with Goldmann Applanation Tonometer. Measurement will be used to categorize each subject as having Low IOP (7 to 16 mmHg), Medium IOP (>16 to <23 mmHg), or High IOP (>23 mmHg).
  Arms: Goldmann Applanation Tonometer
Device: IOP with comparator ORA G3 and ic100 tonometers — Measurement of IOP with Ocular Response Analyzer G3 and ic100 tonometers.
  Arms: ORA G3 and ic100
Device: IOP with Tono-Vera Tonometer — Measurement of IOP with Tono-Vera Tonometer
  Arms: Tono-Vera Tonometer

SUMMARY:
Determine if the Tono-Vera Tonometer accurately measures intraocular pressure (IOP). The hypothesis of this test is to confirm the Tono-Vera Tonometer is equivalent to the Goldmann Applanation Tonometer (within +/- 5.0 mmHg).

DETAILED DESCRIPTION:
The Tono-Vera Tonometer (Reichert, Inc.) is a portable rebound tonometer intended to measure IOP. Subjects will undergo a standard ophthalmologic examination. Subjects will then be measured with four tonometers: Goldmann Applanation Tonometer (C.S.O. SRL), Ocular Response Analyzer G3 (Reichert, Inc.), iCare ic100 tonometer (iCare Finland Oy), and Tono-Vera Tonometer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female, between the ages of 18 and 90 years old;
* Be able and willing to provide signed informed consent
* Be able to follow study instructions

Exclusion Criteria:

* Subjects with only one functional eye;
* Subjects with one eye having poor or eccentric fixation;
* Subjects with central corneal thickness greater than 600 µm or less than 500 µm (about 2 standard deviations the human mean);
* Subjects with corneal scarring or who have had corneal surgery, including corneal laser surgery;
* Subjects with concomitant ocular diseases such as: microphthalmos, buphthalmos, nystagmus, keratoconus, severe dry eye syndrome, blepharospasm, any other corneal or conjunctival pathology or infection;
* Contact lens wearers;
* Known allergy to proparacaine or fluorescein as these are used to anesthetize the eye and allow IOP measurement, respectively, when used with the GAT.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Demonstrate compliance with ANSI Z80.10-2014-Ophthalmics-Ophthalmic Instruments-Tonometers. | Through study completion, approximately 4 months.
  Subjects will be distributed into Low IOP, Medium IOP, and High IOP groups based on Goldmann Applanation Tonometer measurements. The Tono-Vera Tonometer measurements will be within +/-5.0 mmHg of the Goldmann Applanation Tonometer measurements in all groups.

SECONDARY OUTCOMES:
Data collection for two measurement modes. | Through study completion, approximately 4 months.
  Tono-Vera has two measurement modes: A 6-measurement mode & "Quick" measurement mode. The 6-measurement mode will be used during this study. It will be possible to post-process the results to determine the IOP value that would have been obtained using Quick mode. As such the sponsor will be able to ensure the accuracy of both measurement modes compared to Goldmann Tonometry.
Data collection for device calibration. | Through study completion, approximately 4 months.
  The study will collect data on a large number of patients over a wide range of IOP values. The sponsor may use the collected data in a post-hoc analysis to verify that the Tono-Vera Tonometer factory calibration is optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Tseng, MD, PhD, Principal Investigator — Department of Opthalmology, Duke University
Locations (1):
- Department of Ophthalmology, Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No